CLINICAL TRIAL: NCT00970866
Title: Efficacy of Lipid-based Nutrient Supplements (LNS) for Pregnant and Lactating Women and Their Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 223623
Record Dates: First submitted 2009-09-01; First posted 2009-09-03 (Estimated); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Anemia; Malnutrition; Stunting
Keywords: multiple micronutrients; home fortification; complementary foods; infant feeding; lipid-based nutrient supplements
MeSH Terms: conditions — Anemia; Malnutrition; Growth Disorders | interventions — Iron; Folic Acid; Population Groups; Hypoxanthine Phosphoribosyltransferase

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Iron and Folic Acid (IFA) (Active Comparator)
  Interventions: Dietary Supplement: Iron and Folic Acid (IFA); Dietary Supplement: Multiple Micronutrient (MMN) group; Dietary Supplement: Lipid-based Nutrient Supplements (LNS) group
- Multiple Micronutrient (MMN) (Active Comparator)
  Interventions: Dietary Supplement: Iron and Folic Acid (IFA); Dietary Supplement: Multiple Micronutrient (MMN) group; Dietary Supplement: Lipid-based Nutrient Supplements (LNS) group
- Lipid-based Nutrient Supplements (LNS) (Active Comparator)
  Interventions: Dietary Supplement: Iron and Folic Acid (IFA); Dietary Supplement: Multiple Micronutrient (MMN) group; Dietary Supplement: Lipid-based Nutrient Supplements (LNS) group

INTERVENTIONS:
Dietary Supplement: Iron and Folic Acid (IFA) — Pregnant women will receive one (1) Iron (60 mg) and Folic Acid (400 mcg) (IFA) tablet daily during pregnancy, and a tablet containing calcium (Ca) only (akin to a placebo) during lactation; there will be no supplementation for infants born to the women. The Fe/FA tablets will be taken each day with water after meals
Dietary Supplement: Multiple Micronutrient (MMN) group — Pregnant women will receive one (1) Multiple Micronutrient tablet daily during pregnancy and the first 6 months of lactation; there will be no supplementation for infants born to the women. The MMN tablets will be taken each day with water after meals
Dietary Supplement: Lipid-based Nutrient Supplements (LNS) group — Pregnant women will receive 20 g of LNS-P&L daily during pregnancy and the first 6 months of lactation, whilst infants born to the women will receive 20 g of LNS-20gM daily from 6 to 18 mo of age.
  The LNS products (LNS-P&L and LNS-20gM) will be consumed by being added to prepared food (usually mixed with complementary foods, for the child). Mothers will consume the full sachet of LNS (20 g/day) at one meal each day. Dosage and directions for use of the LNS product for children will be as follows: 20 g (~4 teaspoons) per day divided into 2 portions and consumed at two different times of the day (2 x 2 teaspoons). Mix the portion of the supplement to be consumed with 2-3 tablespoons of the already prepared food (as done previously in our study in Ghana (1)), and eat the mixture before eating the rest of the food. Do not cook food with the supplement. Store supplement at room temperature. There is no need for refrigeration.

SUMMARY:
In Ghana, low micronutrient intakes among pregnant women are a major problem. The standard nutritional intervention during pregnancy is iron-folic acid tablets, but adherence is low. The investigators have pioneered the use of multiple micronutrient-fortified semi-solid pastes called Lipid-based Nutrient Supplements (LNS) (made using vegetable oil, groundnut, milk, sugar, and micronutrients), and the investigators' previous studies show that the approach could have great potential for use by pregnant and lactating women.

This study aims to evaluate the effects of LNS-P&L designed for pregnant and lactating women and LNS-20gM designed for infants. Pregnant women (n=864) randomly selected from ante-natal clinics in Yilo and Manya Krobo districts of Ghana will be randomized to receive daily (a) Group 1: Iron/ Folic Acid tablets during pregnancy, and a tablet containing calcium (Ca) only (akin to a placebo) during lactation (6 mo), (b) Group 2: Multiple Micronutrient tablets during pregnancy and the first six months of lactation, or (c) Group 3: LNS-P&L during pregnancy and lactation, whilst their infants receive LNS-20gM daily from 6 to 18 months. There are two primary outcomes namely:

1. Maternal primary outcome: Birth length
2. Child primary outcome: Child length-for-age z-score at 18 mo.

The investigators hypothesize that a) mean birth length and length-for-age at 18 mo will be greater in children whose mothers are in Group 2 than those whose mothers are in Group 1, and b) children whose mothers are in Group 3 will have greater birth length and length-for-age at 18 mo than the children in either of the other two groups.

DETAILED DESCRIPTION:
Introduction:

Inadequate nutrient intakes during pregnancy remain a major problem worldwide. The standard nutritional intervention during pregnancy is iron-folic acid tablets, but adherence is generally quite low. We have pioneered the use of lipid-based nutrient supplements (LNS), which are multiple micronutrient-fortified semi-solid pastes made using vegetable oil, groundnut paste, milk, sugar, and micronutrients, for home fortification of complementary foods for infants. Given results of previous studies with Nutributter in Ghana (1, 2) and similar LNS in Malawi (3, 4) we believe that the food-based approach using LNS has the potential to improve the nutritional status of these women, and thereby also enhance their children's growth and micronutrient status.

Our consortium has formulated LNS-P&L for pregnant and lactating women, and modified the Nutributter for children, which has been called LNS-20gM in this trial. The LNS-20gM provides generally the Recommended Nutrient Intakes (RNI) for 18 vitamins and minerals for infants from 6 to 18 mo of age. The LNS-P&L is modeled on the UNICEF/WHO/UNU international multiple micronutrient preparation (UNIMMAP) for pregnant and lactating women and similar products used in Guinea Bissau (5). Each supplement (20 g/day) will provide 118 kcal/day. Both LNS products (LNS-P&L and LNS-20gM) will, in addition to the multiple micronutrients provided in the MMN, supply energy (118 kcal/d), fat (11 g/d), protein (2.6 g/d), the essential fatty acids linoleic acid (=1.29 g/d) and a-linolenic acid (0.29 to >0.6 g/d), as well as calcium, phosphorus, potassium and magnesium.

Objectives

The study has two objectives, which are:

1. To evaluate the effect of LNS-P&L on the nutritional status of Ghanaian pregnant and lactating women.
2. To assess the effect of LNS-P&L given to pregnant and lactating women and LNS-20gM provided to children from 6 to 18 mo of age on child growth and micronutrient status.

Procedures

1. Recruitment:

   This study will be a community-based, randomized controlled trial with three intervention groups. Potential subjects will be Ghanaian pregnant women attending usual ante-natal clinics at the Government Hospitals at Atua and Akuse, and the St Martins de Porres Catholic Hospital at Agormanya (Manya Krobo District of Ghana), and the Somanya Polyclinic at Somanya (Yilo Krobo District of Ghana).

   Enrolment into the study will be done in two steps. First, pregnant women who meet an initial set of criteria will be asked their consent (sign a Screening Consent Form) to participate in a pre-enrolment screening using a Screening Questionnaire. During this screening, which will be conducted at the clinics, results of the routine ante-natal examination already entered in the Ante-natal Cards will be inspected. The screening questionnaire will also collect additional information, such as description of place of residence, not recorded in the Ante-natal cards.

   Second, women who pass the screening will be contacted in their homes, where we will provide them with additional details of the study and seek their consent for recruitment. If they agree, they will sign a recruitment consent form, and enrolment will be said to be completed. Immediately, we will collect background demographic and socioeconomic information in the home using a Baseline Questionnaire, and schedule the women to come to the laboratory to complete a baseline anthropometric and laboratory assessment (blood and urine sampling, hemoglobin, blood pressure and Ultrasound for gestational age).

   Pregnant women (n = 864) who have completed the baseline assessments and remain eligible for the study will be randomly assigned (using opaque envelopes with group designations) to one of three groups: (1) Group 1: Iron and Folic Acid, (2) Group 2: Multiple Micronutrient (MMN), and (3) Group 3: Lipid-based Nutrient Supplements (LNS).
2. Follow up:

   Pregnant women will be followed-up through delivery, up to 6 mo postpartum (i.e. remaining part of pregnancy from time of recruitment + 6 mo of lactation), the infants born to the women will be followed-up from birth to 18 mo of age. Field Workers will visit subjects in their homes biweekly during pregnancy and weekly from birth to 18 mo to provide supplements and collect data on morbidity and adherence. In the case of multiple births by a woman, (e.g. twins or triplets), one baby will be randomly selected immediately after delivery to be the index child from whom infant data and blood samples will be collected. Anthropometric data will be collected from the unselected twin or triplets, and those in Group 3 will receive LNS-20gM (because of the cultural belief that twins and triplets, etc., must be treated the same), but blood samples will not be collected from the unselected child. In case of loss of child/children during or after delivery, the mother will be followed-up until 6 mo postpartum. In case of loss of mother during or after delivery, the baby will be followed-up until 18 mo of age.

   If any woman in the study is recommended to take additional vitamins and/ or minerals by her physician, we will work with the physician to ensure that any supplement given does not lead to excess intakes.
3. Outcome measures:

The study will have two primary outcomes namely:

1. Maternal primary outcome: Birth length, and
2. Child primary outcome: Child length-for-age z-score at 18 mo.

   Secondary outcomes include:

   i. Maternal:
   * Anthropometric status (weight, BMI, mid upper arm circumference and sub- scapular skin-fold thickness) at ~ 36 wk gestation and at 6, 12, and 18 mo postpartum.
   * Pregnancy outcomes (birth weight, gestational age).
   * Anemia, micronutrient (iron, vitamin A, B-vitamins, zinc) and EFA status, and malarial antigen at ~ 36 wk gestation and 6 mo postpartum.
   * Total plasma cholesterol at ~ 36 wk gestation.
   * Blood pressure and urinary iodine, isoprostane (marker of oxidative stress) and 8-hydroxy-2'deoxyguanosine (8-OHdG) (marker of DNA damage) at 36 wk gestation.
   * Breast milk composition (EFA, vitamin A, B-vitamins, iodine) at 6 mo postpartum.
   * Depressive symptoms (which may be related to EFA status) at 6 mo postpartum.

   ii. Child:
   * Anthropometric status (weight, length, head circumference and mid upper arm circumference) at birth and 3, 6, 12 and 18 mo.
   * Anemia, micronutrient (iron, vitamin A, B-vitamins, iodine) and EFA status, and malarial antigen at 6 and 18 mo.
   * Morbidity between 6 and 18 mo.
   * Child feeding practices and maternal report of child sleep patterns at 6, 12 and 18 mo.
   * Energy intake from complementary foods at 9 and 15 mo.
   * Antibody response to measles vaccination at 12 mo.
   * Achievement of five motor milestones (sitting without support, standing alone, walking with assistance, walking alone and running) and four other developmental milestones (pronouncing single words like mama / dada, waving goodbye, eating by self, drinking from a cup) from 0 to 18 mo.
   * Neuro-behavioral development at 18 mo of age.

   First Post-intervention Follow-up Study: Detailed description

   Introduction:

   Previous research has suggested that nutrition during pregnancy and early childhood can have long term effects on growth, health, and cognition. Only a few studies conducted back in the 1970's, including those in Guatemala (7) and Colombia (8, 9), have followed a cohort that was provided nutrition supplementation during both pregnancy and early childhood. The International Lipid-Based Nutrient Supplements (iLiNS)-DYAD Trial in Ghana examined the effects of a lipid-based nutrient supplement (LNS) provided to women during pregnancy and the first 6 months postpartum, and to their infants from 6 until 18 months of age. Re-assessing the children from that trial at 4-6 years of age is important because this is a critical time for certain longer-term outcomes, such as cognitive development (e.g. school readiness) and body composition prior to puberty.

   Main objective The main objective of this first follow-up study is to evaluate the impact of the iLiNS DYAD-Ghana intervention among participants (women and their children) and their families at 2-4 years post-intervention.

   Primary objectives

   To determine the effects of LNS-P&L given to women during pregnancy and the first 6 mo post-partum, and LNS-20gM given to their children from 6 to 18 months of age on the following outcomes at 4-6 years of age:
   1. Child growth
   2. Child neurobehavioral development

      Secondary objectives:

      To determine the effects of LNS-P&L given to women during pregnancy and the first 6 mo post-partum, and LNS-20gM given to their children from 6 to 18 months of age on the following outcomes at 4-6 years of age:

   a) Health status and stress response of the children b) Sweet taste preferences and food and drink preferences of the children. c) Mental and physical health status of the women after receiving LNS-P&L. d) Caregiver investments in the index child and close siblings. e) Growth of the next younger sibling of the index child. f) Epigenetic DNA modifications of the index child g) Child activity levels

   Study design The study is designed as a follow-up study of a randomized controlled trial. Eligible women and mothers or caregivers of eligible children who took part in the iLiNS DYAD-Ghana intervention trial from 2009 to 2014 will be contacted for enrollment. Fathers and/or younger siblings of eligible children, if available, will also be enrolled.Ethical approval for the study will be obtained from the institutional review boards of the University of California in Davis, the University of Ghana College of Basic and Applied Sciences, and the Ghana Health Service.

   Inclusion criteria
   1. Mothers and children: Participated in the iLiNS DYAD-Ghana trial.
   2. Fathers: Both child and wife (child's mother) participated in the iLiNS DYAD-Ghana trial.

      Exclusion criteria

      Potential participants will be excluded if any of the following is present:

   a) Severe illness or injury which may interfere with data collection, eg. malignancy, etc.

   b) Unwillingness to participate in or cooperate with the study procedures.

   Procedures
   1. Recruitment Eligible mothers and fathers will be contacted in their homes, whereupon their informed consent will be sought for their own participation in the study, and the participation of their children. Where an eligible child lives in the care of a caregiver (instead of a parent or parents), informed consent for the child's participation will be sought from the caregiver and at least one parent, if possible.
   2. Data collection

   Data will be collected at the following contact points:

   i. Four (4) visits by study workers to the homes of participants:
   * Home visit #1: This will occur at or shortly after enrolment. Field workers will collect background socio-economic and demographic information. Enrollment and anthropometric measurement of fathers, as well as anthropometric measurements of younger siblings, may occur at this or any of the subsequent home visits.
   * Home visit #2: Will normally occur within the 7 days after Home visit #1. Study workers will collect children's morbidity data, and arrange with mothers/caregivers to complete the first visit to the central data collection location.
   * Home visit #3: Normally, this will occur within 2 weeks after the Home visit #1. Study worker will: (a) collect mothers'/caregivers' report of their children's taste preference; (b) collect information on the mother's perception of the iLiNS intervention (c) collect saliva samples (sub-set of mothers/index children) to determine cortisol; and, (d) arrange with women (sub-set) to have their children complete the second visit to the central data collection location.
   * Home visit #4: Normally, this will occur within 5 weeks after enrolment. Study workers will administer questionnaires (motor and neurocognitive development questionnaires) and arrange for mother and child to visit the hospital laboratory for more data/sample collection.

   ii. Two (2) visits by mothers and/or children to a central data collection location:

   • Data collection location visit #1: Normally, this will occur between the first and the second week after enrolment. Tasks will include: (a) Anthropometric measurements; (b) Developmental assessments; (c) Deuterium dosing and saliva samples collection for assessment of children's body composition; and (d) Distribution of accelerometers to a sub-sample of children for assessment of physical activity.

   • Data collection location visit #2: Will occur for a sub-set of children normally after 2 weeks following enrollment. These children will complete a sweet taste preference test and a photo game to examine food and drink preference.

   iii. Visit by mothers and children to the Hospital laboratory: Data/sample collection will include: (a) saliva samples (second time for cortisol analysis); (b) mothers' reproductive history; (c) children's clinical examination (Otoscope data); (d) blood pressure; (e) cheek swab; (f) hair sample collection; and (g) blood hemoglobin measurements.

   c. Outcome measures

   Outcome measures will include the following 8 major domains:

1) Growth and body composition of the index child 2) Neurobehavioral development of the index child 3) Health status and stress response of the index child 4) Sweet taste and food/drink preferences of the index child 5) Maternal mental health and stress response 6) Retrospective perceptions of the LNS intervention, and investments" in the index child and close siblings 7) Growth status of the next younger sibling of the index child 8) Activity level of index child 9) Epigenetic effects of the intervention on the index child

Second Post-intervention Follow-up Study: Detailed description

Introduction:

At birth, infants depend completely on their caregivers to regulate their emotional and behavioral states. As the central and autonomic nervous systems develop rapidly during the first two years of life, infants progressively develop self-regulatory skills. These skills lay the foundation for social-emotional skills during childhood and adulthood, which are critical for mental health, success in school and the workplace, and healthy peer and family relationships. Very few studies have examined factors that influence the development of social-emotional regulation in low- and middle-income countries, where an estimated 250 million children are at risk for not fulfilling their developmental potential, partly due to undernutrition. Adequate nutrient intake is essential during pregnancy and infancy, providing the building blocks for nervous system development. In the first follow-up study of the iLiNS-DYAD-G trial in Ghana, receiving LNS predicted fewer social-emotional difficulties at age 4-6 years, and LNS buffered children from the negative effects of materially and socially disadvantaged home environments on social-emotional well-being. Despite these protective effects, overall a high percentage of children had social-emotional difficulty scores in the abnormally high range at age 4-6 years (25% compared to 4-10% in other published studies), suggesting that children in the study area in Ghana are at high risk for the early development of social-emotional difficulties.

Main objective of the second follow-up study:

The main objective of the second follow-up study is to examine the long-term effects of SQ-LNS during pregnancy and infancy on autonomic nervous system regulation and white matter microstructure properties at age 8-12 years, and to determine whether neural effects account for protective effects of LNS on social-emotional functioning at this age, as youths transition into early adolescence, which is a period of high susceptibility to the onset of depressed mood and depressive disorder.

Specific objectives of the second follow-up study:

To determine the effects of LNS-P&L given to women during pregnancy and the first 6 mo post-partum, and LNS-20gM given to their children from 6 to 18 months of age on the following outcomes at 8-12 years of age:

1. Child and adolescent social-emotional development (e.g., SDQ, SCARED, MFQ)
2. Child and adolescent self-regulation (e.g., executive function, risk taking)
3. Child and adolescent autonomic nervous system function
4. Characteristics of child and adolescent brain structure (e.g., white matter microstructure, cortical volume and thickness)
5. Child and adolescent neurobehavioral development (e.g., cognition, literacy and arithmetic)
6. Child and adolescent health and anthropometric status
7. Child and adolescent pubertal development
8. Child and adolescent school performance
9. Maternal cognition and mental health

Study design:

The study is designed as a follow-up study of a randomized controlled trial. Eligible women and mothers or caregivers of eligible children who took part in the iLiNS DYAD-Ghana intervention trial from 2009 to 2014 will be contacted for enrollment. Ethical approval for the study will be obtained from the institutional review boards of the University of California Davis and the Ghana Health Service.

Inclusion criteria:

Mothers and children: Participated in the iLiNS DYAD-Ghana trial.

Exclusion criteria:

Potential participants will be excluded if any of the following is present:

Severe illness or injury which may interfere with data collection, eg. malignancy, etc.

Unwillingness to participate in or cooperate with the study procedures.

Procedures

1. Recruitment Eligible mothers and children will be contacted in their homes, whereupon their informed consent will be sought for their own participation in the study, and the participation of their children. Where an eligible child lives in the care of a caregiver (instead of a parent or parents), informed consent for the child's participation will be sought from the caregiver and at least one parent, if possible.
2. Data collection

Data will be collected at the following contact points:

i. Home visit by study workers to the homes of participants. Field staff will explain the study and obtain informed consent. Consenting participants will be administered a survey to collect demographic and school information (name and location of the child's school and teacher), other caregiver report questionnaires, and assessment of the home environment.

ii. Project office visit. Normally, this will occur between the first and the second week after enrolment. Tasks will include: (a) Autonomic nervous system assessments, (b) Social-emotional and self-regulation assessments, (c) Other neurobehavioral assessments; (d) Anthropometric measurements, (e) Pubertal assessment, (f) blood pressure; (g) hair sample collection; and (h) blood hemoglobin measurements and blood spot collection.

iii. School visit. Field staff will visit the child's school to administer teacher-report questionnaires of the child's behavior.

iv. Visit to hospital for MRI scan (subsample). A subsample of 240 children will be invited to the hospital to participate in a structural MRI scan with a diffusion MRI acquisition.

c. Outcome measures

Outcome measures will include the following major domains:

1. Child and adolescent social-emotional development (e.g., SDQ, SCARED, MFQ)
2. Child and adolescent self-regulation (e.g., executive function, risk taking)
3. Child and adolescent autonomic nervous system function
4. Characteristics of child and adolescent brain structure (e.g., white matter microstructure, cortical volume and thickness)
5. Child and adolescent neurobehavioral development (e.g., cognition, literacy and arithmetic)
6. Child and adolescent health and anthropometric status
7. Child and adolescent pubertal development
8. Child and adolescent school performance
9. Maternal cognition and mental health

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* No more than 20 wk of gestation
* Given Ante-natal Cards of the Ghana Health Service
* Completed the initial routine ante-natal examination at the clinics
* HIV negative or status unknown (as from the Ante-natal card)
* Free from chronic disease e.g. malignancy requiring frequent medical attention (as from the Ante-natal card)
* Residing in the Manya Krobo or Yilo Krobo district
* Prepared to sign an informed consent
* Living in the area throughout the duration of the study
* Acceptance of home visitors

Exclusion Criteria:

* Known asthmatic or history of allergy towards peanut or milk products
* Concurrent participation in another clinical trial
* Severe illness warranting hospital referral

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3499 (Actual)
Dates: Start 2009-11; Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Maternal primary outcome is child length at birth | 0 - 48 hr after birth
Child primary outcome is child length-for-age Z-score (LAZ, based on WHO 2006 growth standards) at 18 months of age | 18 months after birth

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn G. Dewey, PhD, Principal Investigator — UC Davis; Anna Lartey, PhD, Principal Investigator — +233 21 513294; Seth Adu-Afarwuah, PhD, Principal Investigator — University of Ghana; Elizabeth L Prado, PhD, Principal Investigator — University of California, Davis
Locations (4):
- Ghana (4):
  - St. Martin de Porre's Hospital, Agomanya
  - Atua Government Hospital, Atua
  - Kpong Reproductive and Child Health (RCH) Center, Kpong
  - Somanya Polyclinic, Somanya

REFERENCES:
- [Background] Adu-Afarwuah S, Lartey A, Brown KH, Zlotkin S, Briend A, Dewey KG. Randomized comparison of 3 types of micronutrient supplements for home fortification of complementary foods in Ghana: effects on growth and motor development. Am J Clin Nutr. 2007 Aug;86(2):412-20. doi: 10.1093/ajcn/86.2.412. PMID 17684213
- [Background] Adu-Afarwuah S, Lartey A, Brown KH, Zlotkin S, Briend A, Dewey KG. Home fortification of complementary foods with micronutrient supplements is well accepted and has positive effects on infant iron status in Ghana. Am J Clin Nutr. 2008 Apr;87(4):929-38. doi: 10.1093/ajcn/87.4.929. PMID 18400716
- [Background] Phuka JC, Maleta K, Thakwalakwa C, Cheung YB, Briend A, Manary MJ, Ashorn P. Postintervention growth of Malawian children who received 12-mo dietary complementation with a lipid-based nutrient supplement or maize-soy flour. Am J Clin Nutr. 2009 Jan;89(1):382-90. doi: 10.3945/ajcn.2008.26483. Epub 2008 Dec 3. PMID 19056572
- [Background] Phuka JC, Maleta K, Thakwalakwa C, Cheung YB, Briend A, Manary MJ, Ashorn P. Complementary feeding with fortified spread and incidence of severe stunting in 6- to 18-month-old rural Malawians. Arch Pediatr Adolesc Med. 2008 Jul;162(7):619-26. doi: 10.1001/archpedi.162.7.619. PMID 18606932
- [Background] Kaestel P, Michaelsen KF, Aaby P, Friis H. Effects of prenatal multimicronutrient supplements on birth weight and perinatal mortality: a randomised, controlled trial in Guinea-Bissau. Eur J Clin Nutr. 2005 Sep;59(9):1081-9. doi: 10.1038/sj.ejcn.1602215. PMID 16015266
- [Background] Rivera JA, Martorell R, Ruel MT, Habicht JP, Haas JD. Nutritional supplementation during the preschool years influences body size and composition of Guatemalan adolescents. J Nutr. 1995 Apr;125(4 Suppl):1068S-1077S. doi: 10.1093/jn/125.suppl_4.1068S. PMID 7722709
- [Background] Mora JO, de Paredes B, Wagner M, de Navarro L, Suescun J, Christiansen N, Herrera MG. Nutritional supplementation and the outcome of pregnancy. I. Birth weight. Am J Clin Nutr. 1979 Feb;32(2):455-62. doi: 10.1093/ajcn/32.2.455. PMID 420135
- [Background] Super CM, Herrera MG, Mora JO. Long-term effects of food supplementation and psychosocial intervention on the physical growth of Colombian infants at risk of malnutrition. Child Dev. 1990 Feb;61(1):29-49. PMID 2307045
- [Derived] Partington LC, Yuan H, Demuyakor ME, Adu-Afarwuah S, Guyer AE, Dewey KG, Kumordzie SM, Oaks BM, Arnold CD, Prado EL, Hastings PD. Early-life nutritional supplementation protects against home environmental risks in Ghanaian children's social-emotional development. Front Nutr. 2025 Aug 20;12:1571677. doi: 10.3389/fnut.2025.1571677. eCollection 2025. PMID 40909891
- [Derived] Nti H, Adu-Afarwuah S, Oaks BM, Prado EL, Arnold CD, Hastings PD, Guyer AE, Dewey KG, Amponsah B, Bentil HJ, Mensah MO, Adjetey E, Tan X, Aryee LMD, Labi FBA, Manu A. Impact of Small-Quantity Lipid-Based Nutrient Supplements on Pubertal Status of 9-13-Year Olds: A Follow-Up Study of the iLiNS-DYAD-Ghana Trial. Curr Dev Nutr. 2024 Sep 26;8(12):104458. doi: 10.1016/j.cdnut.2024.104458. eCollection 2024 Dec. PMID 39758592
- [Derived] Aryee LMD, Adu-Afarwuah S, Prado EL, Guyer AE, Arnold CD, Dewey KG, Amponsah B, Manu A, Oaks BM, Bentil HJ, Nti H, Ayete Labi FB, Mensah MO, Adjetey E, Hastings PD. Effect of Early-Life Lipid-Based Nutrient Supplement and Home Environment on Autonomic Nervous System Regulation at 9-11 Years: A Follow-Up of a Randomized Controlled Trial. Matern Child Nutr. 2025 Apr;21(2):e13789. doi: 10.1111/mcn.13789. Epub 2024 Dec 16. PMID 39679749
- [Derived] Bentil HJ, Adu-Afarwuah S, Prado EL, Arnold CD, Hastings PD, Guyer AE, Mensah MO, Manu A, Tan X, Adjetey E, Amponsah B, Demuyakor ME, Dewey KG, Oaks BM. Sustained effects of small-quantity lipid-based nutrient supplements provided during the first 1000 days on child growth at 9-11 y in a randomized controlled trial in Ghana. Am J Clin Nutr. 2024 Feb;119(2):425-432. doi: 10.1016/j.ajcnut.2023.10.033. Epub 2023 Dec 29. PMID 38309829
- [Derived] Hong BV, Zheng JJ, Romo EZ, Agus JK, Tang X, Arnold CD, Adu-Afarwuah S, Lartey A, Okronipa H, Dewey KG, Zivkovic AM. Seasonal Factors Are Associated with Activities of Enzymes Involved in High-Density Lipoprotein Metabolism among Pregnant Females in Ghana. Curr Dev Nutr. 2023 Nov 23;7(12):102041. doi: 10.1016/j.cdnut.2023.102041. eCollection 2023 Dec. PMID 38130330
- [Derived] Prado EL, Adu-Afarwuah S, Arnold CD, Adjetey E, Amponsah B, Bentil H, Dewey KG, Guyer AE, Manu A, Mensah M, Oaks BM, Ocansey M, Tan X, Hastings PD. Prenatal and postnatal small-quantity lipid-based nutrient supplements and children's social-emotional difficulties at ages 9-11 y in Ghana: follow-up of a randomized controlled trial. Am J Clin Nutr. 2023 Aug;118(2):433-442. doi: 10.1016/j.ajcnut.2023.05.025. Epub 2023 May 29. PMID 37257564
- [Derived] Adu-Afarwuah S, Arnold CD, Lartey A, Okronipa H, Maleta K, Ashorn P, Ashorn U, Dewey KG. Prevalence of morbidity symptoms among pregnant and postpartum women receiving different nutrient supplements in Ghana and Malawi: A secondary outcome analysis of two randomised controlled trials. Matern Child Nutr. 2023 Jul;19(3):e13501. doi: 10.1111/mcn.13501. Epub 2023 Apr 6. PMID 37021807
- [Derived] Hong BV, Zhu C, Wong M, Sacchi R, Rhodes CH, Kang JW, Arnold CD, Adu-Afarwuah S, Lartey A, Oaks BM, Lebrilla CB, Dewey KG, Zivkovic AM. Lipid-Based Nutrient Supplementation Increases High-Density Lipoprotein (HDL) Cholesterol Efflux Capacity and Is Associated with Changes in the HDL Glycoproteome in Children. ACS Omega. 2021 Nov 18;6(47):32022-32031. doi: 10.1021/acsomega.1c04811. eCollection 2021 Nov 30. PMID 34870025
- [Derived] Adu-Afarwuah S, Arnold CD, Lartey A, Okronipa H, Maleta K, Ashorn P, Ashorn U, Fan YM, Matchado A, Kortekangas E, Oaks BM, Jackson KH, Dewey KG. Small-Quantity Lipid-Based Nutrient Supplements Increase Infants' Plasma Essential Fatty Acid Levels in Ghana and Malawi: A Secondary Outcome Analysis of the iLiNS-DYAD Randomized Trials. J Nutr. 2022 Jan 11;152(1):286-301. doi: 10.1093/jn/nxab329. PMID 34543432
- [Derived] Abreu AM, Young RR, Buchanan A, Lofgren IE, Okronipa HET, Lartey A, Ashorn P, Adu-Afarwuah S, Dewey KG, Oaks BM. Maternal Blood Pressure in Relation to Prenatal Lipid-Based Nutrient Supplementation and Adverse Birth Outcomes in a Ghanaian Cohort: A Randomized Controlled Trial and Cohort Analysis. J Nutr. 2021 Jun 1;151(6):1637-1645. doi: 10.1093/jn/nxab018. PMID 33704494
- [Derived] Oaks BM, Adu-Afarwuah S, Kumordzie S, Laudenslager ML, Smith DL, Lin J, Young RR, Arnold CD, Bentil H, Okronipa H, Ocansey M, Dewey KG. Impact of a nutritional supplement during gestation and early childhood on child salivary cortisol, hair cortisol, and telomere length at 4-6 years of age: a follow-up of a randomized controlled trial. Stress. 2020 Sep;23(5):597-606. doi: 10.1080/10253890.2020.1728528. Epub 2020 Feb 24. PMID 32063089
- [Derived] Adu-Afarwuah S, Young RR, Lartey A, Okronipa H, Ashorn P, Ashorn U, Oaks BM, Dewey KG. Supplementation with Small-Quantity Lipid-Based Nutrient Supplements Does Not Increase Child Morbidity in a Semiurban Setting in Ghana: A Secondary Outcome Noninferiority Analysis of the International Lipid-Based Nutrient Supplements (iLiNS)-DYAD Randomized Controlled Trial. J Nutr. 2020 Feb 1;150(2):382-393. doi: 10.1093/jn/nxz243. PMID 31603205
- [Derived] Kumordzie SM, Okronipa H, Arimond M, Adu-Afarwuah S, Ocansey ME, Young RR, Bentil HJ, Tamakloe SM, Oaks BM, Dewey KG. Maternal and child factors associated with child body fatness in a Ghanaian cohort. Public Health Nutr. 2020 Feb;23(2):309-318. doi: 10.1017/S1368980019001745. Epub 2019 Jul 25. PMID 31340880
- [Derived] Kumordzie SM, Adu-Afarwuah S, Arimond M, Young RR, Adom T, Boatin R, Ocansey ME, Okronipa H, Prado EL, Oaks BM, Dewey KG. Maternal and Infant Lipid-Based Nutritional Supplementation Increases Height of Ghanaian Children at 4-6 Years Only if the Mother Was Not Overweight Before Conception. J Nutr. 2019 May 1;149(5):847-855. doi: 10.1093/jn/nxz005. PMID 31034033
- [Derived] Okronipa H, Arimond M, Arnold CD, Young RR, Adu-Afarwuah S, Tamakloe SM, Ocansey ME, Kumordzie SM, Oaks BM, Mennella JA, Dewey KG. Exposure to a slightly sweet lipid-based nutrient supplement during early life does not increase the level of sweet taste most preferred among 4- to 6-year-old Ghanaian children: follow-up of a randomized controlled trial. Am J Clin Nutr. 2019 Apr 1;109(4):1224-1232. doi: 10.1093/ajcn/nqy352. PMID 30915467
- [Derived] Okronipa H, Arimond M, Young RR, Arnold CD, Adu-Afarwuah S, Tamakloe SM, Bentil HJ, Ocansey ME, Kumordzie SM, Oaks BM, Dewey KG. Exposure to a Slightly Sweet Lipid-Based Nutrient Supplement During Early Life Does Not Increase the Preference for or Consumption of Sweet Foods and Beverages by 4-6-y-Old Ghanaian Preschool Children: Follow-up of a Randomized Controlled Trial. J Nutr. 2019 Mar 1;149(3):532-541. doi: 10.1093/jn/nxy293. PMID 30770539
- [Derived] Kumordzie SM, Adu-Afarwuah S, Young RR, Oaks BM, Tamakloe SM, Ocansey ME, Okronipa H, Prado EL, Dewey KG. Maternal-Infant Supplementation with Small-Quantity Lipid-Based Nutrient Supplements Does Not Affect Child Blood Pressure at 4-6 Y in Ghana: Follow-up of a Randomized Trial. J Nutr. 2019 Mar 1;149(3):522-531. doi: 10.1093/jn/nxy285. PMID 30753625
- [Derived] Ocansey ME, Adu-Afarwuah S, Kumordzie SM, Okronipa H, Young RR, Tamakloe SM, Oaks BM, Dewey KG, Prado EL. Prenatal and postnatal lipid-based nutrient supplementation and cognitive, social-emotional, and motor function in preschool-aged children in Ghana: a follow-up of a randomized controlled trial. Am J Clin Nutr. 2019 Feb 1;109(2):322-334. doi: 10.1093/ajcn/nqy303. PMID 30721937
- [Derived] Oaks BM, Jorgensen JM, Baldiviez LM, Adu-Afarwuah S, Maleta K, Okronipa H, Sadalaki J, Lartey A, Ashorn P, Ashorn U, Vosti S, Allen LH, Dewey KG. Prenatal Iron Deficiency and Replete Iron Status Are Associated with Adverse Birth Outcomes, but Associations Differ in Ghana and Malawi. J Nutr. 2019 Mar 1;149(3):513-521. doi: 10.1093/jn/nxy278. PMID 30629202
- [Derived] Adu-Afarwuah S, Young RT, Lartey A, Okronipa H, Ashorn P, Ashorn U, Oaks BM, Arimond M, Dewey KG. Maternal and Infant Supplementation with Small-Quantity Lipid-Based Nutrient Supplements Increases Infants' Iron Status at 18 Months of Age in a Semiurban Setting in Ghana: A Secondary Outcome Analysis of the iLiNS-DYAD Randomized Controlled Trial. J Nutr. 2019 Jan 1;149(1):149-158. doi: 10.1093/jn/nxy225. PMID 30624674
- [Derived] Adams KP, Ayifah E, Phiri TE, Mridha MK, Adu-Afarwuah S, Arimond M, Arnold CD, Cummins J, Hussain S, Kumwenda C, Matias SL, Ashorn U, Lartey A, Maleta KM, Vosti SA, Dewey KG. Maternal and Child Supplementation with Lipid-Based Nutrient Supplements, but Not Child Supplementation Alone, Decreases Self-Reported Household Food Insecurity in Some Settings. J Nutr. 2017 Dec;147(12):2309-2318. doi: 10.3945/jn.117.257386. Epub 2017 Oct 4. PMID 28978680
- [Derived] Okronipa H, Adu-Afarwuah S, Lartey A, Ashorn P, Vosti SA, Young RR, Dewey KG. Maternal supplementation with small-quantity lipid-based nutrient supplements during pregnancy and lactation does not reduce depressive symptoms at 6 months postpartum in Ghanaian women: a randomized controlled trial. Arch Womens Ment Health. 2018 Feb;21(1):55-63. doi: 10.1007/s00737-017-0752-7. Epub 2017 Jul 11. PMID 28698916
- [Derived] Adu-Afarwuah S, Lartey A, Okronipa H, Ashorn P, Ashorn U, Zeilani M, Arimond M, Vosti SA, Dewey KG. Maternal Supplementation with Small-Quantity Lipid-Based Nutrient Supplements Compared with Multiple Micronutrients, but Not with Iron and Folic Acid, Reduces the Prevalence of Low Gestational Weight Gain in Semi-Urban Ghana: A Randomized Controlled Trial. J Nutr. 2017 Apr;147(4):697-705. doi: 10.3945/jn.116.242909. Epub 2017 Mar 8. PMID 28275100
- [Derived] Oaks BM, Young RR, Adu-Afarwuah S, Ashorn U, Jackson KH, Lartey A, Maleta K, Okronipa H, Sadalaki J, Baldiviez LM, Shahab-Ferdows S, Ashorn P, Dewey KG. Effects of a lipid-based nutrient supplement during pregnancy and lactation on maternal plasma fatty acid status and lipid profile: Results of two randomized controlled trials. Prostaglandins Leukot Essent Fatty Acids. 2017 Feb;117:28-35. doi: 10.1016/j.plefa.2017.01.007. Epub 2017 Jan 25. PMID 28237085
- [Derived] Klevor MK, Adu-Afarwuah S, Ashorn P, Arimond M, Dewey KG, Lartey A, Maleta K, Phiri N, Pyykko J, Zeilani M, Ashorn U. A mixed method study exploring adherence to and acceptability of small quantity lipid-based nutrient supplements (SQ-LNS) among pregnant and lactating women in Ghana and Malawi. BMC Pregnancy Childbirth. 2016 Aug 30;16(1):253. doi: 10.1186/s12884-016-1039-0. PMID 27577112
- [Derived] Adu-Afarwuah S, Lartey A, Okronipa H, Ashorn P, Peerson JM, Arimond M, Ashorn U, Zeilani M, Vosti S, Dewey KG. Small-quantity, lipid-based nutrient supplements provided to women during pregnancy and 6 mo postpartum and to their infants from 6 mo of age increase the mean attained length of 18-mo-old children in semi-urban Ghana: a randomized controlled trial. Am J Clin Nutr. 2016 Sep;104(3):797-808. doi: 10.3945/ajcn.116.134692. Epub 2016 Aug 17. PMID 27534634
- [Derived] Prado EL, Abbeddou S, Adu-Afarwuah S, Arimond M, Ashorn P, Ashorn U, Brown KH, Hess SY, Lartey A, Maleta K, Ocansey E, Ouedraogo JB, Phuka J, Some JW, Vosti SA, Yakes Jimenez E, Dewey KG. Linear Growth and Child Development in Burkina Faso, Ghana, and Malawi. Pediatrics. 2016 Aug;138(2):e20154698. doi: 10.1542/peds.2015-4698. PMID 27474016
- [Derived] Prado EL, Adu-Afarwuah S, Lartey A, Ocansey M, Ashorn P, Vosti SA, Dewey KG. Effects of pre- and post-natal lipid-based nutrient supplements on infant development in a randomized trial in Ghana. Early Hum Dev. 2016 Aug;99:43-51. doi: 10.1016/j.earlhumdev.2016.05.011. Epub 2016 Jul 6. PMID 27391572
- [Derived] Adu-Afarwuah S, Lartey A, Okronipa H, Ashorn P, Zeilani M, Baldiviez LM, Oaks BM, Vosti S, Dewey KG. Impact of small-quantity lipid-based nutrient supplement on hemoglobin, iron status and biomarkers of inflammation in pregnant Ghanaian women. Matern Child Nutr. 2017 Apr;13(2):e12262. doi: 10.1111/mcn.12262. Epub 2016 Feb 29. PMID 26924599
- [Derived] Oaks BM, Laugero KD, Stewart CP, Adu-Afarwuah S, Lartey A, Ashorn P, Vosti SA, Dewey KG. Late-Pregnancy Salivary Cortisol Concentrations of Ghanaian Women Participating in a Randomized Controlled Trial of Prenatal Lipid-Based Nutrient Supplements. J Nutr. 2016 Feb;146(2):343-52. doi: 10.3945/jn.115.219576. Epub 2016 Jan 13. PMID 26764321
- [Derived] Klevor MK, Haskell MJ, Lartey A, Adu-Afarwuah S, Zeilani M, Dewey KG. Lipid-Based Nutrient Supplements Providing Approximately the Recommended Daily Intake of Vitamin A Do Not Increase Breast Milk Retinol Concentrations among Ghanaian Women. J Nutr. 2016 Feb;146(2):335-42. doi: 10.3945/jn.115.217786. Epub 2016 Jan 6. PMID 26740682
- [Derived] Adu-Afarwuah S, Lartey A, Okronipa H, Ashorn P, Zeilani M, Peerson JM, Arimond M, Vosti S, Dewey KG. Lipid-based nutrient supplement increases the birth size of infants of primiparous women in Ghana. Am J Clin Nutr. 2015 Apr;101(4):835-46. doi: 10.3945/ajcn.114.091546. Epub 2015 Feb 11. PMID 25833980